CLINICAL TRIAL: NCT00680680
Title: Phase 4 Study of Dual Five Alpha Reductase Inhibition Combined With Alpha Blockade in Men With Refractory Urinary Retention Secondary to BPH
Brief Title: Treatment of Refractory Urinary Retention Secondary to Benign Prostatic Hyperplasia (BPH) With Dual Five Alpha Reductase Inhibition Combined With an Alpha Blocker
Acronym: AUR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Franklin D. Gaylis, MD Inc. (Other)
Responsible Party: Franklin D. Gaylis, M.D., MEDRESEARCH
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUR
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Urinary Retention; Benign Prostatic Hyperplasia
Keywords: Urinary retention secondary to benign prostatic hyperplasia
MeSH Terms: conditions — Urinary Retention; Prostatic Hyperplasia | interventions — Dutasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Dutasteride — Patients will continue on their alpha blocker in addition to Dutasteride 0.5mg daily for a maximum of 3 months

SUMMARY:
To determine whether the addition of a dual Five Alpha Reductase Inhitor (Dutasteride) will alleviate urinary retention secondary to BPH in who have failed a voiding trial without a catheter. Following treatment with an Alpha Blocker alone.

ELIGIBILITY:
Inclusion Criteria:

1. Males betewen the ages of 50 and 90 years of age.Written informed consent.
2. Men with acute urinary retention attributed to bladder outlet obstruction caused by BPH, who have failed atleast 1 week trial of alpha blocker treatment.
3. PSA level equal to or greater than 1.5ng/ml and equal to or less than 15 ng/ml.

Exclusion Criteria:

1. Urinary retention attributed to a neurogenic or myogenic bladder dysfunction.
2. Use of psychotrophic medications.
3. Use of antichollinergic medications.
4. Prostate cancer.
5. Allery to five alpha reductase inhibitors.
6. Prior prostate surgery.
7. Urethral stricture.
8. Bladder calculi.
9. Invasive bladder cancer.
10. Inability to understand or agree with the requirements of the study.
11. Any investigational drug received within 30 days prior of study entry.

Ages: 50 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2004-05; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franklin D Gaylis, MD, Principal Investigator — Director/Sponsor